CLINICAL TRIAL: NCT01148992
Title: Phase 1, Double-Blind, Placebo-Controlled Assessment of Potential Interactions Between Intravenous Cocaine and Lofexidine
Brief Title: Interactions Between Intravenous (IV) Cocaine and Lofexidine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lofexidine-0001
Record Dates: First submitted 2010-06-17; First posted 2010-06-23 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-08

CONDITIONS: Cocaine Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — lofexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lofexidine (Active Comparator)
  Interventions: Drug: Lofexidine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lofexidine — 0.8mg alone and concurrent with IV cocaine infusions of 20 mg and 40 mg
  Arms: Lofexidine
Drug: Placebo — 0mg
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess potential interactions between intravenous (IV) cocaine and treatment with lofexidine.

DETAILED DESCRIPTION:
To determine the safety of daily oral lofexidine alone and concurrent with IV cocaine infusions of 20 mg and 40 mg in cocaine-experienced, non-opiate-addicted volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Be volunteers who meet Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria for cocaine abuse or dependence and are non-treatment seeking at the time of the study.
* Be between 18 and 50 years of age, inclusive.
* Be currently use cocaine. Use must be confirmed by a positive urine test for cocaine metabolites once within the outpatient screening period.
* Be able to verbalize understanding of the consent form and provide written informed consent.
* Females must have a negative pregnancy test within 72 hours prior to receiving the first infusion of cocaine. They must also be postmenopausal, have had a hysterectomy, been sterilized, or agree to use one of the following methods of birth control:

  * diaphragm and condom by partner
  * intrauterine device (that does not contain progesterone) and condom by partner
  * sponge and condom by partner
  * complete abstinence from sexual intercourse

Note: Oral contraceptives, Depo-Provera, Norplant, Patch, and intrauterine progesterone contraceptive system are not allowed.

Exclusion Criteria:

* Please contact site for more information

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Adverse Event and Cardiovascular Response | Daily, up to 9 days
  Adverse Events will measured during follow-up at weeks 14-21

SECONDARY OUTCOMES:
Pharmacokinetics (PK) Parameter of Cocaine and Benzoylecgonine (BE) | Daily, up to 9 days
PK of Lofexidine | Daily, up to 9 days
Visual Analog Scale (VAS) | Daily, up to 9 days
Brief Substance Abuse Craving Scale (BSCA) | Daily, up to 9 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No